CLINICAL TRIAL: NCT04810195
Title: Early neo2 Registry of the Acurate neo2 TAVI Prosthesis
Status: Completed | Type: Observational
Sponsor: Andreas Rück (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor-Investigator, Andreas Rück, Principal Investigator, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Other Study IDs: HKN AR01
Record Dates: First submitted 2021-03-07; First posted 2021-03-22 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Aortic Valve Stenosis
Keywords: TAVR
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Boston Scientific Acurate neo2 TAVR device — The newest generation of the Acurate neo2 TAVR device, launched in Europe in 2020.

SUMMARY:
The Early neo2 registry will study up to 500 patients treated with the updated Boston Acurate neo2 TAVI prosthesis at various European hospitals. The data is gathered from routine healthcare and there are no study-mandated additional procedures. The main endpoint is a combined efficiency and safety endpoint after 30 days. Imaging data (echocardiography, computed tomography and aortography) will be analysed centrally by a core lab.

DETAILED DESCRIPTION:
Background and rationale The Boston Scientific Acurate neo2 TAVI prosthesis was launched commercially in Europe in September 2020 as a successor to the original Acurate neo prosthesis. Modifications include an added sealing skirt. The original Acurate neo failed to reach non-inferiority to other TAVI prostheses in two randomized trials. There is a need to gather initial safety and efficacy data from this next generation prosthesis, as there is no larger dataset presented after the CE-mark study of the Acurate neo2.

Project objectives To gather initial safety and efficacy data in the initial up to 500 consecutive patients treated with the Acurate neo2 in various European sites.

Karolinska will be the coordinating center for data collection.

Methods Data will be collected in an anonymous form and sent to Karolinska for compilation and statistics. Data collection will continue until 500 patients are reached (April, 2021).

Statistics Standard descriptive statistics will be used for the main results. For the comparison to SCOPE data (with the original Acurate neo prosthesis) on postoperative aortic insufficiency, standard statistical methods will used (Fishers exact test for categorical variables, and t-test for continuous measurements such as amount of regurgitation by videodensitometry).

Core lab studies The core lab analyses will be performed at CORRIB in Galway (Prof. Serruys et al).

ELIGIBILITY:
Inclusion Criteria:

* that a Acurate neo2 prosthesis has been inserted into the sheath (i.e. a procedure has been started).

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The first 500 consecutive patients treated with the Acurate neo2 from up to 15 European sites which have started using the Acurate neo2.
Sampling Method: Probability Sample
Enrollment: 554 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
MACE | 30 days
  any of
  * Postoperative aortic insuffiency moderate or higher (in hospital echo, site reported)
  * Postoperative new permanent pacemaker (in hospital)
  * 30 days mortality
  * 30 days stroke
  * Acute Kidney Injury (AKIN grade 3) (in hospital)

SECONDARY OUTCOMES:
Rate of Postoperative aortic insufficiency more than mild by transthoracic echo | Within 7 days of procedure
  Core-lab analysis of the postoperative transthoracic echo for aortic insufficiency: percentage of patients with more than mild insufficiency
Rate of Postoperative aortic insufficiency more than mild by aortography | Same day as procedure
  Core-lab analysis of the aortogram in the end of the procedure for quantification of aortic insufficiency (videodensitometry): rate of patients with more than mild insuffiency
Postoperative aortic valve gradients | Within 7 days of procedure
  Aortic prosthesis mean gradient (mmHg) on postoperative transthoracic echocardiogram
Rate of major acute procedural complications | Same day as procedure
  Intraprocedural complications such as valve embolization, need for second valve, anular rupture
Procedural contrast use | Same day as procedure
  The average amount of contrast in ml per procedure

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Rück, MD PhD, Principal Investigator — Karolinska University Hospital
Locations (4):
- Rigshospitalet, Copenhagen, Denmark
- Kerckhoff Klinik, Bad Nauheim, Germany
- Sweden (2):
  - Lund University Hospital, Lund
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided